CLINICAL TRIAL: NCT05880173
Title: SCREaning of Advanced Liver Fibrosis Using Non-Invasive Tests in General Population
Acronym: SCREANIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 49RC22_0399
Record Dates: First submitted 2023-01-06; First posted 2023-05-30 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Screening; Advanced Liver Fibrosis
Keywords: Screening; advanced liver fibrosis; non-invasive tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic FIB4 (Other): Only one arm because diagnostic study evaluating blood test using elastometry and liver biopsy as reference
  Interventions: Diagnostic Test: FIB4

INTERVENTIONS:
Diagnostic Test: FIB4 — Diagnostic procedure :
  FIB4 blood tests in medical analysis laboratories. If FIB4 positive, Non invasive spacialized evaluation (transient elastography and FibroMeter) by a specialist and if necessery liver biopsy, endoscopy and/or echography

SUMMARY:
The main objective of the study is to evaluate the pertinence of initiating screening for advanced hepatic fibrosis after a FIB4 result > 2.67 automatically calculated in the local laboratory and followed by a specialized hepatic evaluation.

DETAILED DESCRIPTION:
Chronic liver diseases are insidious diseases characterized by inflammation of the liver parenchyma responsible for a progressive accumulation of fibrosis until cirrhosis and hepatocellular carcinoma (HCC). Cirrhosis and HCC are respectively the 11th and 16th most frequent causes of death in the world, and are responsible for 2 million deaths each year. Cirrhosis and HCC are most often diagnosed too late with a median survival of 18-24 months.

The degree of hepatic fibrosis is the main predictive factor of the risk of hepatic complications (decompensation of cirrhosis, HCC) in chronic liver diseases.

Hepatic fibrosis is described in 5 stages from F0 (no fibrosis) to F4 (cirrhosis). It is well accepted that patients with advanced hepatic fibrosis (F3 and F4) are at the highest risk of developing complications of cirrhosis and/or HCC. It is therefore necessary to identify these patients in order to offer them specialized management.

Tests have been developed over the last two decades for the non-invasive diagnosis of liver fibrosis, essentially the fibrosis blood test (FIB4) and liver elastometry devices (fibroScan). The FIB4 is a simple blood test that is easy to calculate from the usual inexpensive blood parameters (ASAT, ALAT, platelets). The recommendations of French, European and American scientific societies are unanimous and recommend targeted screening for liver fibrosis in patients with hepatic risk factors using FIB4 as a first line test.

To facilitate screening by general practitioners, several French consortia of medical analysis laboratories have set up routine calculation of FIB4 on all biological tests, including platelets, AST and ALT, without regard to the patient's risk factors for liver disease. This approach is not in concordance with the recommendations of the scientific societies (targeted screening in patients with hepatic risk factors) and needs to be evaluated.

The purpose of this study is to evaluate if the procedure for diagnosing hepatic fibrosis implemented by some local laboratories and based on an automated calculation of FIB4 is pertinent.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* Blood sample taken at a medical testing laboratory selected for the study.
* Biology without high risk of false positive result for FIB4 (AST and ALT ≤ 300 IU/l ; Platelets ≥ 50 G/l and < 500 G/l.)
* FIB4 > 2.67 after automatic calculation in the medical laboratory less than 3 months old
* Signature of informed consent to participate in the study

Exclusion Criteria:

* Ongoing specialized follow-up for a chronic liver disease
* Difficulty understanding the French language
* Pregnant women, breastfeeding or parturient women
* Persons suspended from liberty by judicial or administrative decision
* Persons under legal protection
* Persons unable to express their consent
* Non affiliation to a social security system

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of advanced hepatic fibrosis. | 3 months maximum
  The endpoint for this objective will be the diagnosis of advanced liver fibrosis is a stage of F3-4 fibrosis on liver biopsy (NASH-CRN classification), in patients with a FIB4> 2.67 and a FibroScan result ≥ 8 kPa.

SECONDARY OUTCOMES:
Determine the rate of patients requiring second-line evaluation by elastometry | 3 months maximum
  The endpoint for this objective will be the rate of patients with FIB4 >2.67.
Determine the rate of patients requiring management by a liver disease specialist. | 3 months maximum
  The endpoint for this objective will be the rate of patients with a FIB4 >2.67 and then a FibroScan ≥8.0 kPa.
Determine the average cost spent on a patient diagnosed with advanced liver fibrosis | 3 months maximum
  The endpoint for this objective will be the average direct cost of all procedures performed in the screening procedure.
Determine patient adherence to the screening procedure | 3 months maximum
  The endpoint for this objective will be the rate of patients performing the procedures in accordance with the screening procedure.
Determine risk factors associated with advanced liver fibrosis, and consequently the subgroup of patients for whom screening should be a priority | 3 months maximum
  The endpoint for this objective will be multivariate analysis of risk factors according to the stage of detected liver fibrosis
Determine the rate of patients with a significant liver complication in the population of patients with risk factors | 3 months maximum
  The endpoints for this objective will be the number of diagnosed hepatocellular carcinoma and esophageal/gastric varices with bleeding risk.

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Chu Angers, Angers
  - Chu Bordeaux, Angers
  - Chu Grenoble Alpes, Grenoble
  - Centre Hospitalier de Lens, Lens
  - Hopital Saint Joseph, Marseille
  - Chu Nancy, Nancy

IPD SHARING:
Plan to Share IPD: No